CLINICAL TRIAL: NCT03668600
Title: An Open-label, Long-term Extended Access Protocol for Rapastinel as Adjunctive or Monotherapy Treatment in Patients With Major Depressive Disorder
Brief Title: Study of Adjunctive or Monotherapy Rapastinel Treatment in Patients With Major Depressive Disorder (MDD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision to stop the program
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAP-MD-99
Record Dates: First submitted 2018-08-28; First posted 2018-09-12 (Actual); Results first posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Depressive Disorder, Major
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — GLYX-13 peptide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rapastinel (Experimental): Rapastinel 450 mg (prefilled syringe, weekly or biweekly or up to 4 weeks at the investigator's discretion intravenous IV administration)
  Interventions: Drug: Rapastinel

INTERVENTIONS:
Drug: Rapastinel — Rapastinel 450 mg (prefilled syringe, weekly or biweekly or up to 4 weeks at the investigator's discretion intravenous IV administration)

SUMMARY:
Multicenter, open-label, long-term extended access treatment protocol in adult patients with a primary diagnosis of MDD.

ELIGIBILITY:
Inclusion Criteria:

* Completion of lead-in study
* Adequate therapeutic benefit in the lead-in study to justify continuation of treatment with rapastinel in the judgement of the investigator

Exclusion Criteria:

* Suicide risk, as determined by meeting any of the following criteria:

  1. A suicide attempt within the past year
  2. Significant risk, as judged by the investigator, based on the psychiatric interview or information collected in the Columbia- Suicide Severity Rating Scale (C-SSRS) at any visit in the lead-in study
  3. Montgomery-Asberg Depression Rating Scale (MADRS) Item 10 score ≥ 5 at any visit during participation in the lead-in study where MADRS was conducted.
* At imminent risk of injuring self or others or causing significant damage to property, as judged by the investigator
* Females who are pregnant, breastfeeding, or planning to become pregnant or breastfeed during participation
* Females of childbearing potential and male partners of females of childbearing potential, not using a reliable means of contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hoogerheyde, Study Director — Allergan
Locations (74):
- United States (74):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Harmonex Neuroscience Research, Dothan, Alabama
  - NoesisPharma, Phoenix, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - California Pharmaceutical Research Institute, Inc, Anaheim, California
  - Southern California Research LLC., Beverly Hills, California
  - ATP Clinical Research Inc., Costa Mesa, California
  - ProScience Research Group, Culver City, California
  - Pharmacology Research Institute, Encino, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Sun Valley Research Center, Imperial, California
  - Irvine Center for Clinical Research, Inc, Irvine, California
  - Synergy Clinical Research Center of Escondido, Lemon Grove, California
  - Pharmacology Research Institute, Los Alamitos, California
  - CITrials, Riverside, California
  - California Neuroscience Research, Sherman Oaks, California
  - Viking Clinical Research, Temecula, California
  - Pacific Clinical Research Medical, Upland, California
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Reliable Clinical Research, Hialeah, Florida
  - Meridien Research, Lakeland, Florida
  - Innovative Clinical Research, Inc, Lauderhill, Florida
  - Research Centers of America, Oakland Park, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - David A. Medina, MD, Orlando, Florida
  - Institute for Advanced Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Attalla Consultants, LLC, Smyrna, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR - Baber Research, Inc., Naperville, Illinois
  - University of Kansas School of Medicine Clinical Trial Unit, Wichita, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Louisiana Clinical Research, Shreveport, Louisiana
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - Coastal Research Associates, South Weymouth, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Healthy Perspectives - Innovative Mental Health Services. PLLC, Nashua, New Hampshire
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Neuroscience, Inc, Albuquerque, New Mexico
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Patient Priority Clinical Sites, Cincinnati, Ohio
  - The Ohio State University Department of Psychiatry, Columbus, Ohio
  - Midwest Clinical Research Center LLC, Dayton, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - Red River Medical Research Center, LLC, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Inc, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Summit Research Network LLC, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Dr. Cherian Verghese, Norristown, Pennsylvania
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Donald J. Garcia, Jr., MD, PA, Austin, Texas
  - Community Clinical Research, Austin, Texas
  - Houston Clinical Trials, Bellaire, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Earle Research, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Psychiatric and Behavioral Solutions, Salt Lake City, Utah
  - Psychiatric Alliance of the Blue Ridge, Inc, Charlottesville, Virginia

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from RAP-MD-99, completed 1 of the rapastinel lead-in studies - RAP-MD-04, RAP-MD-05, RAP-MD-06 or RAP-MD-33.
Period: Overall Study
Arm/Group | Rapastinel
Started | 230
Completed | 0
Not Completed | 230
Not completed — Study Terminated by the Sponsor | 157
Not completed — Protocol Violation | 1
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 56
Not completed — Lack of Efficacy | 7
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The Open-label Safety Population will consist of all participants who signed the RAP-MD-99 ICF and who received at least 1 dose of open-label rapastinel during the OLTP of the protocol.
Arm/Group | Rapastinel
Number analyzed (Participants) | 230
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 209
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 200
  More than one race | 2
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 84.70 (18.55)
Height [Median (Standard Deviation); unit: cm] | 166.22 (8.82)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.63 (6.66)

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Experiencing One or More Treatment Emergent Adverse Events (TEAEs)
Description: A Treatment Emergent Adverse Event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. An Adverse Drug Reaction was a harmful and unintended reaction that is incurred during routine administration or use of the drug, whose causal relationship with the drug cannot be excluded.
Time Frame: Up to 45 Weeks
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Rapastinel
Number analyzed (Participants) | 230
Participants | 100

ADVERSE EVENTS:
Time Frame: Up to 45 Weeks
Description: The Open-label Safety Population will consist of all participants who signed the RAP-MD-99 ICF and who received at least 1 dose of open-label rapastinel during the OLTP of the protocol.
Arm/Group | Rapastinel
All-Cause Mortality (participants affected / at risk) | 0/230
Serious Adverse Events (participants affected / at risk) | 4/230
Other Adverse Events (participants affected / at risk) | 14/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Rapastinel (N=230)
Ventricular tachycardia (Cardiac disorders) | 1
Device malfunction (Product Issues) | 1
Pericardial effusion (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/191
Rib fracture (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rapastinel (N=230)
Dysgeusia (Nervous system disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT03668600/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT03668600/SAP_001.pdf